CLINICAL TRIAL: NCT06902779
Title: Enhanced Collaboration Between Hospital and Community Pharmacists to Improve the Hospital Discharge Process
Brief Title: Evaluation of the Impact of a Collaboration Between Hospital and Community Pharmacists at Hospital Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacie des Hopitaux de l'Est Lemanique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ECHOPHARM
Record Dates: First submitted 2025-03-11; First posted 2025-03-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Polypharmacy
Keywords: transition of care; pharmacists; hospital discharge; collaboration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Participants in the control arm will benefit from the usual standard of care currently provided in routine clinical practice. Physicians performs medication reconciliation on their own and hand-out the prescription to the patient the day of discharge. The patient then goes to the pharmacy for a classical drug dispensation.
- Intervention arm (Experimental): Participants in the intervention group will benefit from the hospital pharmacist's support to optimize medication management and ensure a safe and effective discharge process.
  Interventions: Other: Support of the hospital pharmacist for the medication management at hospital discharge

INTERVENTIONS:
Other: Support of the hospital pharmacist for the medication management at hospital discharge — 1) The hospital pharmacist calls the community pharmacy the day before discharge to order unusual or specific medications 2) The day of discharge, the hospital pharmacist performs a medication reconciliation in collaboration with the hospital physician 3) Once completed, the discharge prescription is sent to the community pharmacy before the patient is discharged. 4) The hospital pharmacist calls the community pharmacy to provide additional information about the patient and the prescription and to answer any questions. Additional information will help the community pharmacist to understand the prescription : administrative data, clinical data, medication-related information, patient follow-up and patient concerns.
  Arms: Intervention arm

SUMMARY:
The aim of this study is to evaluate the impact of an enhanced collaboration between a hospital pharmacist and a community pharmacist during hospital discharge. For patients taking multiple medications, hospitalization often involves numerous changes to their treatment regimen. For community pharmacies, discharge prescriptions are often complex, and they sometimes lack the information that pharmacists need to deliver the treatment as safely as possible. As a result, there is a risk of medication errors, and a risk for patients. We aim to evaluate the benefits of this collaboration for adult patients admitted to the internal medicine ward of a regional hospital who are taking seven or more drugs and are being discharged to home.

The main question it aims to answer is : Does the enhanced collaboration reduce the number of drug-related problems encountered by community pharmacists with discharge prescriptions ? Researchers will compare patients when a hospital pharmacist is involved during the discharge process and when he or she is not involved, which corresponds to normal care.

The hospital pharmacist will not perform the intervention directly on the patient, but only with the community pharmacy. Once they agree to participate in the study, patients will only have to go to their usual community pharmacy after discharge and accept that the hospital transmits medical information to their usual pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the internal medicine ward for more than 48 hours
* Patients prescribed seven or more drugs at the time of screening
* Patients discharged to home
* Patients able to give informed consent as documented by signature

Exclusion Criteria:

* Patient discharged to another hospital, nursing home or rehabilitation clinic
* Refusal of the community pharmacy to participate
* Inability to sign consent and follow the procedures of the study, due to language problems, psychological disorders, dementia, alterations of consciousness and lack of judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of drug-related problems on the hospital discharge prescription | 7 days after hospital discharge
  Community pharmacists will assess the number of drug-related problems (DRP) on the discharge that they faced when preparing the discharge medication. They will have to use the PharmDISC system, which is a validated tool for referencing drug-related problems faced in the community which was adapted from the drug-related problems classification system of the Pharmaceutical Care Network Europe (PCNE). Community pharmacists will also document the intervention performed for each DRP, and the resolution (yes/no) of the DRP.

SECONDARY OUTCOMES:
Patient's satisfaction | 7 days after hospital discharge
  Patients' satisfaction related to their visit at the pharmacy after hospital discharge will be assessed using a questionnaire. Patients will be contacted via email or telephone
Community pharmacists' satisfaction | Through study completion, approximately 6 months
  The satisfaction of community pharmacists with the service provided by the hospital pharmacist at patient discharge will be evaluated
30 day readmission rate | 30 days after hospital discharge
  Number of participants with hospital emergency department visits and hospital readmission in the same hospital within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Blanc, PharmD, PhD, Study Director — Pharmacie des Hôpitaux de l'Est Lémanique
Locations (1):
- Hôpital Riviera-Chablais, Vaud-Valais, Rennaz, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared includes demographic and study outcomes, with a data summary Data will be anonymized and shared in a secure format (CSV)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD data will be available 6 months after publication of the first study results and for 10 years
Access Criteria: Data will be accessible to external researchers, regulatory bodies, and authorized entities under the following conditions:
  Formal request submission detailing the project and data usage. Access granted if the request meets ethical, scientific, and confidentiality criteria.

REFERENCES:
- [Background] Michel B, Hemery M, Rybarczyk-Vigouret MC, Wehrle P, Beck M. Drug-dispensing problems community pharmacists face when patients are discharged from hospitals: a study about 537 prescriptions in Alsace. Int J Qual Health Care. 2016 Dec 1;28(6):779-784. doi: 10.1093/intqhc/mzw111. PMID 27655792
- [Background] Braund R, Coulter CV, Bodington AJ, Giles LM, Greig AM, Heaslip LJ, Marshall BJ. Drug related problems identified by community pharmacists on hospital discharge prescriptions in New Zealand. Int J Clin Pharm. 2014 Jun;36(3):498-502. doi: 10.1007/s11096-014-9935-8. Epub 2014 Apr 4. PMID 24700340
- [Background] Imfeld-Isenegger TL, Studer H, Ceppi MG, Rosen C, Bodmer M, Beeler PE, Boeni F, Haring AP, Hersberger KE, Lampert ML. Detection and resolution of drug-related problems at hospital discharge focusing on information availability - a retrospective analysis. Z Evid Fortbild Qual Gesundhwes. 2021 Nov;166:18-26. doi: 10.1016/j.zefq.2021.08.004. Epub 2021 Sep 15. PMID 34538579
- [Background] Ahmad A, Mast MR, Nijpels G, Elders PJ, Dekker JM, Hugtenburg JG. Identification of drug-related problems of elderly patients discharged from hospital. Patient Prefer Adherence. 2014 Feb 4;8:155-65. doi: 10.2147/PPA.S48357. eCollection 2014. PMID 24523581
- [Background] Maes KA, Studer H, Berger J, Hersberger KE, Lampert ML. Documentation of pharmaceutical care: Validation of an intervention oriented classification system. J Eval Clin Pract. 2017 Dec;23(6):1425-1432. doi: 10.1111/jep.12817. Epub 2017 Sep 29. PMID 28960678
- [Background] Mekonnen AB, McLachlan AJ, Brien JA. Pharmacy-led medication reconciliation programmes at hospital transitions: a systematic review and meta-analysis. J Clin Pharm Ther. 2016 Apr;41(2):128-44. doi: 10.1111/jcpt.12364. Epub 2016 Feb 23. PMID 26913812
- [Background] McCarthy LM, Li S, Fernandes O, Cameron K, Lui P, Wong G, Pariser P, Farrell J, Luke MJ, Guilcher SJT. Enhanced communication between inpatient and community pharmacists to optimize medication management during transitions of care. J Am Pharm Assoc (2003). 2019 Jan-Feb;59(1):79-86.e1. doi: 10.1016/j.japh.2018.09.006. Epub 2018 Nov 13. PMID 30446423
- [Background] Bruhwiler LD, Hersberger KE, Lutters M. Hospital discharge: What are the problems, information needs and objectives of community pharmacists? A mixed method approach. Pharm Pract (Granada). 2017 Jul-Sep;15(3):1046. doi: 10.18549/PharmPract.2017.03.1046. Epub 2017 Aug 25. PMID 28943987
- [Background] Grandchamp S, Blanc AL, Roussel M, Tagan D, Sautebin A, Dobrinas-Bonazzi M, Widmer N. Pharmaceutical Interventions on Hospital Discharge Prescriptions: Prospective Observational Study Highlighting Challenges for Community Pharmacists. Drugs Real World Outcomes. 2022 Jun;9(2):253-261. doi: 10.1007/s40801-021-00288-x. Epub 2021 Dec 31. PMID 34971408
- [Background] Redmond P, Grimes TC, McDonnell R, Boland F, Hughes C, Fahey T. Impact of medication reconciliation for improving transitions of care. Cochrane Database Syst Rev. 2018 Aug 23;8(8):CD010791. doi: 10.1002/14651858.CD010791.pub2. PMID 30136718
- [Background] Ensing HT, Stuijt CC, van den Bemt BJ, van Dooren AA, Karapinar-Carkit F, Koster ES, Bouvy ML. Identifying the Optimal Role for Pharmacists in Care Transitions: A Systematic Review. J Manag Care Spec Pharm. 2015 Aug;21(8):614-36. doi: 10.18553/jmcp.2015.21.8.614. PMID 26233535
- [Background] Mekonnen AB, McLachlan AJ, Brien JA. Effectiveness of pharmacist-led medication reconciliation programmes on clinical outcomes at hospital transitions: a systematic review and meta-analysis. BMJ Open. 2016 Feb 23;6(2):e010003. doi: 10.1136/bmjopen-2015-010003. PMID 26908524
- [Background] Villeneuve Y, Courtemanche F, Firoozi F, Gilbert S, Desbiens MP, Desjardins A, Dinh C, LeBlanc VC, Attia A. Impact of pharmacist interventions during transition of care in older adults to reduce the use of healthcare services: A scoping review. Res Social Adm Pharm. 2021 Aug;17(8):1361-1372. doi: 10.1016/j.sapharm.2020.11.006. Epub 2020 Nov 13. PMID 33250364
- [Background] Banholzer S, Dunkelmann L, Haschke M, Derungs A, Exadaktylos A, Krahenbuhl S, Liakoni E. Retrospective analysis of adverse drug reactions leading to short-term emergency hospital readmission. Swiss Med Wkly. 2021 Jan 20;151:w20400. doi: 10.4414/smw.2021.20400. eCollection 2021 Jan 18. PMID 33516159
- [Background] Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med. 2003 Feb 4;138(3):161-7. doi: 10.7326/0003-4819-138-3-200302040-00007. PMID 12558354